CLINICAL TRIAL: NCT05349994
Title: Extended Physiotherapy After Intensive Care Unit (ICU) Stay: A Prospective Before and After Study
Brief Title: Extended Physiotherapy After Intensive Care Unit (ICU) Stay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Katinka Siesage, RPT, Clinical Specialist Physiotherapist Intensive Care, MSc, Stockholm South General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Improvement project AFE
Record Dates: First submitted 2022-04-13; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Critical Illness; Physical Disability
Keywords: Physical therapy; Physical function
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: The study design was a before and after study. A control group was included for three months and received standard care. An intervention group was then included for six months and received extended amount of physical therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard amount of physical therapy at surgical wards in an urban hospital, corresponding to 1.75 physiotherapy employment on weekdays divided on four wards with a total of approx. 40-48 patients.
- Intervention (Experimental): Extended physiotherapy with an extra 0.5 employment on weekdays, leading to 1-2 physiotherapy session per day for the study participants in the intervention group.
  Interventions: Other: Extended physiotherapy

INTERVENTIONS:
Other: Extended physiotherapy — At admission to the surgical ward after ICU care, participants received an individual rehabilitation plan developed in collaboration with the participants and the ward-based physiotherapist. The rehabilitation plan included specified exercises for 1- 2 sessions of approximately 30 minutes a day. For example breathing exercises, practicing transfer in and out of bed and from sitting to standing, stairclimbing, and walking with or without walking aids.
  Arms: Intervention

SUMMARY:
Patients in an Intensive Care Unit (ICU) are at great risk of muscle atrophy and neuromuscular complications, that could lead to respiratory complications, decreased physical functioning and deteriorated health related quality of life. The objective is to investigate if extended physical therapy in a general ward could lead to increased physical functioning for post-ICU patients.The study hypothesis is that extended physical therapy would lead to increased physical function at hospital discharge compared to standard amount of physical therapy.

DETAILED DESCRIPTION:
The study design is a before and after study. A control group was included for three months and received standard amount of physical therapy at surgical wards, corresponding to 1.75 employment. An intervention group was then included for six months and received extended amount of physical therapy corresponding to an extra 0.5 employment for study participants (2-4 patients/day). The primary outcome was physical function measured with the Chelsea Critical Care Physical Assessment Tool (CPAx), in the ICU and the surgical ward.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* ICU stay >48 hours
* Understand the Swedish language

Exclusion Criteria:

• Patients palliative care with no intention of rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
Changes in physical function according to Chelsea Critical Care Physical Assessment tool (CPAx) | Through study completion, an average of 2 weeks per participant
  Measures physical function in critically ill patients

SECONDARY OUTCOMES:
Feasibility of intervention | Through study completion, an average of 2 weeks per participant
  Number of planned interventions not delivered, and number of safety events.
Length of stay at the ward | Through study completion, an average of 2 weeks per participant
  Number of days at the hospital ward after ICU discharge
Readmission to ICU | Through study completion, an average of 2 weeks per participant
  Number of readmissions to ICU from ward, within each study group

CONTACTS AND LOCATIONS:
Overall Officials: Katinka Siesage, Principal Investigator — Stockholm South General Hospital; Eva Alm- Joelsson, Principal Investigator — Stockholm South General Hospital
Locations (1):
- Stockholm South General Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Data available on request due to privacy/ethical restrictions.